CLINICAL TRIAL: NCT03755323
Title: Establishment of a Database of Patients Suffering From Obesity With a Medical Treatment in the Framework of The Specialized Obesity Center Languedoc-Roussillon CHU Montpellier
Brief Title: Establishment of a Database of Patients Suffering From Obesity With a Medical Treatment
Acronym: Elodie Cohort
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL18_0322
Record Dates: First submitted 2018-11-26; First posted 2018-11-27 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: BMI Greater Than 30
Keywords: Obesity; Nutrition Disorders
MeSH Terms: conditions — Obesity; Nutrition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Obesity is a public health problem, given its prevalence (15% in France in 2012, Obépi survey) but also by the complications that it generates. We were firstly, intersted in bone mineral density during obesity.

We were able to confirm in an observational study that BMD (Z-score)was augmented. We also showed, for the first time, that this increase in Z-score was dependent on sex, severity of obesity and age but also bone site. If the increase in BMD at the level of the bearing zones seems logically to be explained by the hypothesis that the mechanical stresses have an osteogenic effect on the bone tissue, the latter can not in any way respond to the concomitant increase in BMD at non-bearing areas such as the radius.These results suggest that changes in certain systemic compounds induced by obesity may interfere with bone metabolism. recent data also suggest a change in the concentration of pro-glucagon peptides (GLP-1, glicentin, glucagon, etc.) in obese subjects and in bariatric surgery). Although body composition and its variation after surgery could be largely involved in the modification of these peptides, no data on these potential relationships is currently available. However, no data are available for baseline body composition and weight loss data. Finally, 80% of obesity is associated with insulin resistance, a key mechanism in the pathophysiology of type 2 diabetes. A metabolically healthy obesity phenotype is described, although the definition criteria are not consensual.The evolution of this phenotype with aging and with the duration of evolution of obesity is not well described.

Our goal is to create a database of weight-bearing patients in the care setting and to determine the "hormonal dialogue" between peripheral (muscular and adipose) and bone tissues, which may be associated with changes in body composition during obesity and aging, and that according to sex.

ELIGIBILITY:
Inclusion criteria:

- obese patients age above 18 years old

Exclusion criteria:

- non agreement of inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects older than 18 years (BMI greater than 30). These patients are seen in consultation with a request for weight management carried out in the cade care , in the framework of The Specialized Obesity Center Languedoc-Roussillon CHU Montpellier
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
identify the determinants of body composition | 1 day
  Compile a comprehensive database of all patients who are weight-bearing as part of the care to identify the determinants of body composition (lean mass, bone mass, muscle mass) in the obese subject according to sex and age, and the link with the complications of obesity.

SECONDARY OUTCOMES:
Measured plasma concentration | 1 day
  Measured plasma concentration of myokines, adipokines, markers of bone remodeling, incretin-glucagon
measurement of muscle strength | 1 day
  the measurement of muscle strength by hand-grip and performance by 6-minute walk test.

CONTACTS AND LOCATIONS:
Overall Officials: Ariane SULTAN, PR, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC